CLINICAL TRIAL: NCT06271239
Title: Effect of Multicomponent Exercises on the Intrinsic Functional Capacity of Older Adults
Brief Title: Effect of Multicomponent Exercises VIVIFRAIL® in Older Adults
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Pontificia Universidade Católica do Rio Grande do Sul (Other)
Collaborators: Coordenação de Aperfeiçoamento de Pessoal de Nível Superior. (Other Government)
Responsible Party: Principal Investigator, Ângelo José Gonçalves Bós, Full Professor at school of medicine, Pontificia Universidade Católica do Rio Grande do Sul
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: U1111-1299-9167; 65318722.0.0000.5336 (Other: IRB-Pontifical Catholic University of Rio Grande do Sul); RBR-2tq2jky (Other: The Brazilian Registry of Clinical Trials (ReBEC))
Record Dates: First submitted 2024-01-24; First posted 2024-02-21 (Actual); Last update posted 2024-06-06 (Actual); Status verified 2024-06

CONDITIONS: Frailty; Aging; Physical Disability
Keywords: Aging; Public Health; Frailty; Exercise
MeSH Terms: conditions — Frailty; Motor Activity

STUDY DESIGN:
Intervention Model Description: In the Intervention Group (ViviFrail), participants will perform a six-month VIVIFRAIL® protocol-based exercise, adapted to their clinical profile.
  The Group Suggestions for a Healthy Life (CG) will receive exercise suggestions and guidance for maintaining a healthy routine for three months. After, they will undergo a three-month intervention using the VIVIFRAIL® protocol.
  Sample size determination was based on Casas-Herrero et al. (2022). The study assessed the impact of multicomponent training on intrinsic functional capacity, utilizing the Short Physical Performance Battery (SPPB) to gauge balance, gait speed, and lower limb strength on a 0 to 12 scale. Control group: -0.33±1.60 point difference; Treatment group: 1.07±1.52 point difference.
  Considering a 5% alpha and 80% power, 20 participants per group are required. Anticipating a 25% dropout rate, as observed by Tiecker (2021), we plan to enroll 25 participants per group.
Who Masked: Outcomes Assessor
Masking Description: The assessments will be conducted by trained researchers
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group (ViviFrail) (Experimental): Intervention Group: 25 participants will be guided to perform one of the home-based exercise programs from the VIVIFRAIL® protocol, tailored to their clinical conditions and functional capacity.
  Interventions: Other: Intervention group (ViviFrail)
- Group Suggestions for a Healthy Life (CG) (Active Comparator): The control group, also consisting of 25 participants, will receive exercise suggestions and guidance on maintaining a healthy routine for three months. Subsequently, the participants will undergo the intervention with the VIVIFRAIL® program for three months.
  Interventions: Other: Group Suggestions for a Healthy Life (CG)

INTERVENTIONS:
Other: Intervention group (ViviFrail) — The participant will be guided to follow a daily exercise routine at home, lasting 30-45 minutes, from Monday to Friday, over six months. A one-week break every six weeks for reassessment, totaling seven months of activities, will be provided. They will be informed that every six weeks, they may receive new exercises in their exercise passport or continue with the same, based on their physical reassessment. Each exercise passport will have a wheel illustrating the exercise circuit for easy reference. An 'Activity Diary' will be provided for tracking progress and frequency. During 'CIRCUIT' sessions, participants should complete the entire circuit, while 'WALKING' sessions should focus solely on walking for that day. They will be motivated to keep this diary updated. The ViviFrail exercise passports cater to various levels of physical frailty and fall risk and can be accessed at https://vivifrail.com/en/materials-2/.
  Arms: Intervention group (ViviFrail)
Other: Group Suggestions for a Healthy Life (CG) — The participants in the group Suggestions for a healthy life (CG) will receive guidance on maintaining a healthy and independent lifestyle for three months. They will also be provided with a booklet containing strength, balance, and flexibility activities, suggesting that participants perform these activities five times a week, for around 30 minutes per day. At the end of the initial three complete months of the intervention (14 weeks), participants in the control group will commence the ViviFrail exercise protocol and will continue until the end of the study. Throughout the entire study period, participants in the control group will receive the same monitoring as the intervention group.
  Arms: Group Suggestions for a Healthy Life (CG)

SUMMARY:
This study employs a randomized, controlled, paired, single-blind clinical trial design. The targeted demographic comprises individuals aged 60 and above. Following the initial assessment, participants will be randomly allocated to two groups: the Intervention Group (ViviFrail) and the Group Suggestions for a Healthy Life (CG), maintaining a 1:1 allocation ratio. Both the ViviFrail group and CG group will exhibit homogeneity in terms of their clinical characteristics and functional performance. The allocation of participants into respective groups will remain concealed from all assessors, ensuring a single-blind approach.

In the intervention group (ViviFrail), 25 participants will be instructed to engage in tailored physical exercises outlined in the VIVIFRAIL® protocol within the confines of their homes, with adaptations made according to their clinical conditions and functional performance.

Conversely, the Group Suggestions for a Healthy Life (CG) comprising 25 participants will receive exercise suggestions and guidance to maintain a healthy routine for a duration of three months. Subsequently, participants in the CG will undergo the VIVIFRAIL® program intervention for an additional three months.

DETAILED DESCRIPTION:
Objective: This study aims to assess the impact of a multicomponent physical exercise intervention on the intrinsic functional capacity of older adults. Methodology: A randomized, controlled, paired, single-blind clinical trial will be conducted. Participants, aged 60 years or older, will be randomly assigned to either the Intervention Group (ViviFrail) or the Group Suggestions for a Healthy Life (CG). The study sample will consist of older individuals, both men and women, enrolled in the senior groups of the social assistance program administered by the City Hall of Porto Alegre.

The initial assessment will be conducted by outcome evaluators utilizing a set of study instruments, including functionality questionnaires for Activities of Daily Living and Instrumental Activities of Daily Living, Short Physical Performance Battery for evaluating intrinsic functional capacity (focusing on lower limb strength, balance, and gait speed), fall risk assessment, self-perceived health, adverse health outcomes, and a multiprofessional evaluation.

Following the initial assessment, participants meeting the inclusion and exclusion criteria will be randomly allocated to the research groups (ViviFrail and CG). Participants in the ViviFrail group will be categorized based on their functional performance, and the most suitable multicomponent exercise passport from the VIVIFRAIL® protocol will be assigned. The training period will span six months, with reassessments every six weeks and a one-week interval for evaluation, resulting in a total duration of seven months.

Participants in the ViviFrail group will be instructed to perform home exercises five times a week, with each session lasting 30 to 45 minutes. The researcher will provide exercise passports and facilitate familiarization with the proposed training during weekly meetings at locations designated by the social assistance program in Porto Alegre, or through regular phone contact for monitoring purposes.

The CG group will function as the control group, receiving exercise suggestions and guidance on maintaining a healthy routine for three months. Subsequently, they will undergo the VIVIFRAIL® program intervention for an additional three months. The follow-up period will be identical for both groups, with each engaging in eight months of activities.

ELIGIBILITY:
Inclusion Criteria:

* Eligible participants are older adults of both genders, aged at least 60 years.
* Participants must be actively participating in regular meetings of elderly groups within the social assistance program in Porto Alegre.
* Participants should not have severe visual, hearing, or cognitive impairments that could impede the safe completion of proposed assessments or exercises

Exclusion Criteria:

* Participants with scheduled surgeries or procedures within the next eight months hindering engagement in the exercise program are excluded.
* Those unable to sit unsupported for at least 10 minutes during the functional assessment or demonstrating an inability to respond to verbal commands in the cognitive assessment are excluded.
* Exclusion criteria specific to the VIVIFRAIL® exercise protocol include:
* Recent acute myocardial infarction or unstable angina within 6 months
* History of uncontrolled arrhythmias
* Dissecting aortic aneurysm
* Severe aortic stenosis
* Acute endocarditis/pericarditis
* Uncontrolled hypertension
* Acute thromboembolic disease
* Severe acute heart failure
* Severe acute respiratory failure
* Uncontrolled orthostatic hypotension
* Acute decompensation of diabetes mellitus or uncontrolled hypoglycemia
* Recent fracture within the last month
* Any other circumstances deemed prohibitive or risky for engaging in physical activity are also grounds for exclusion.

Min Age: 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2024-05-28 (Actual); Primary Completion 2025-01-31 (Estimated); Study Completion 2025-05-30 (Estimated)

PRIMARY OUTCOMES:
Short physical performance battery | through study completion, an average of 1 year
  It's expected to observe an improvement in intrinsic functional capacity from baseline (start of intervention) to the end of the six-month intervention, as evaluated by the Short physical performance battery. This assessment combines balance, gait speed, and lower limb strength into a single score ranging from 0 (worst) to 12 (best). A clinically significant change will be considered as a 1-point change on the Short physical performance battery.

SECONDARY OUTCOMES:
Barthel Index | through study completion, an average of 1 year
  It is expected to observe improvement in basic activities of daily living (ADL), assessed through the Barthel Index (<20 total dependence; 20-35 severe dependence; 40-55 moderate dependence; ≥60 mild dependence; 100 Independent).
ICOPE questionnaire | through study completion, an average of 1 year
  It is expected to observe improvement in basic activities of daily living (ADL), assessed through the Integrated care for older people (ICOPE) Functional Ability questionnaire (21 points: independent).
Lawton Scale | through study completion, an average of 1 year
  Improvement is expected to be observed in instrumental activities of daily living (IADL), assessed through the Lawton Scale (27 points: independent)
4-meter gait speed | through study completion, an average of 1 year
  An improvement in walking time in the 4-meter gait speed test is expected, where a change of 0.1 m/s is considered clinically relevant.
Five Times Sit-to-Stand | through study completion, an average of 1 year
  Improvement in the performance of the Five Times Sit-to-Stand Test is expected. Good performance will be considered if the participant completes it in ≤14.8 seconds, and poor performance if it's >14.8 seconds.
Balance test in three positions | through study completion, an average of 1 year
  Improvement in balance (0 to 4 points) is expected, determined through tests involving standing with one foot in front of the other, in a semi-tandem position, and in a tandem position. A change of 1 point in the test will be considered an improvement in balance.
Self-perceived health | through study completion, an average of 1 year
  It's expected to observe a change in self-perceived health ("very poor", "poor", "fair", "good", and "excellent")
Adverse health outcomes - falls | through study completion, an average of 1 year
  It's expected to observe changes in adverse health outcomes: falls in the "last three months" ("Yes"; "No")
Adverse health outcomes - hospitalization | through study completion, an average of 1 year
  It's expected to observe changes in adverse health outcomes: hospitalization in the "last three months" ("Yes"; "No")
Adverse health outcomes - institutionalization | through study completion, an average of 1 year
  It's expected to observe changes in adverse health outcomes: institutionalization in the "last three months" ("Yes"; "No")

CONTACTS AND LOCATIONS:
Overall Officials: Angelo Bós, Phd, Principal Investigator — Pontificia Universidade Católica do Rio Grande do Sul
Locations (4):
- Brazil (4):
  - Industrial Retirement and Pension Institute (IAPI), Porto Alegre, Rio Grande do Sul
  - The First of May Community Center (CEPRIMA), Porto Alegre, Rio Grande do Sul
  - The Older Adult Day Center (CDI), Porto Alegre, Rio Grande do Sul
  - The Vila Floresta Community Center (CECOFLOR), Porto Alegre, Rio Grande do Sul

IPD SHARING:
Plan to Share IPD: Yes
Each participant will be assigned a sequential Arabic number for identification. In all databases shared with individuals not directly involved in the research, these numbers will be used as identifiers, replacing personal information such as parts of the name, address, phone numbers, and names of family members/caregivers.
  All data will be available for five years to any readers of the article interested in conducting secondary analyses, provided they submit a proposal that does not compromise the authors' future publication interests. Requests should be sent to the corresponding author via email, and the data will be made available in an Excel spreadsheet.
  Additional documents will be available for five years from the publication date, including the study protocol and the data request form.
Supporting Information: Study Protocol, ICF
Time Frame: five years
Access Criteria: Send an email to the research lead

REFERENCES:
- [Background] Casas-Herrero A, Saez de Asteasu ML, Anton-Rodrigo I, Sanchez-Sanchez JL, Montero-Odasso M, Marin-Epelde I, Ramon-Espinoza F, Zambom-Ferraresi F, Petidier-Torregrosa R, Elexpuru-Estomba J, Alvarez-Bustos A, Galbete A, Martinez-Velilla N, Izquierdo M. Effects of Vivifrail multicomponent intervention on functional capacity: a multicentre, randomized controlled trial. J Cachexia Sarcopenia Muscle. 2022 Apr;13(2):884-893. doi: 10.1002/jcsm.12925. Epub 2022 Feb 11. PMID 35150086
- [Background] Casas-Herrero A, Anton-Rodrigo I, Zambom-Ferraresi F, Saez de Asteasu ML, Martinez-Velilla N, Elexpuru-Estomba J, Marin-Epelde I, Ramon-Espinoza F, Petidier-Torregrosa R, Sanchez-Sanchez JL, Ibanez B, Izquierdo M. Effect of a multicomponent exercise programme (VIVIFRAIL) on functional capacity in frail community elders with cognitive decline: study protocol for a randomized multicentre control trial. Trials. 2019 Jun 17;20(1):362. doi: 10.1186/s13063-019-3426-0. PMID 31208471
- [Background] Cadore EL, Casas-Herrero A, Zambom-Ferraresi F, Idoate F, Millor N, Gomez M, Rodriguez-Manas L, Izquierdo M. Multicomponent exercises including muscle power training enhance muscle mass, power output, and functional outcomes in institutionalized frail nonagenarians. Age (Dordr). 2014 Apr;36(2):773-85. doi: 10.1007/s11357-013-9586-z. Epub 2013 Sep 13. PMID 24030238
- [Background] Martinez-Velilla N, Casas-Herrero A, Zambom-Ferraresi F, Suarez N, Alonso-Renedo J, Contin KC, de Asteasu ML, Echeverria NF, Lazaro MG, Izquierdo M. Functional and cognitive impairment prevention through early physical activity for geriatric hospitalized patients: study protocol for a randomized controlled trial. BMC Geriatr. 2015 Sep 15;15:112. doi: 10.1186/s12877-015-0109-x. PMID 26374430
- [Background] Sanchez-Sanchez JL, de Souto Barreto P, Anton-Rodrigo I, Ramon-Espinoza F, Marin-Epelde I, Sanchez-Latorre M, Moral-Cuesta D, Casas-Herrero A. Effects of a 12-week Vivifrail exercise program on intrinsic capacity among frail cognitively impaired community-dwelling older adults: secondary analysis of a multicentre randomised clinical trial. Age Ageing. 2022 Dec 5;51(12):afac303. doi: 10.1093/ageing/afac303. PMID 36580558
- [Background] Courel-Ibanez J, Buendia-Romero A, Pallares JG, Garcia-Conesa S, Martinez-Cava A, Izquierdo M. Impact of Tailored Multicomponent Exercise for Preventing Weakness and Falls on Nursing Home Residents' Functional Capacity. J Am Med Dir Assoc. 2022 Jan;23(1):98-104.e3. doi: 10.1016/j.jamda.2021.05.037. Epub 2021 Jun 29. PMID 34197791
- [Background] Kis O, Buch A, Stern N, Moran DS. Minimally supervised home-based resistance training and muscle function in older adults: A meta-analysis. Arch Gerontol Geriatr. 2019 Sep-Oct;84:103909. doi: 10.1016/j.archger.2019.103909. Epub 2019 Jul 8. PMID 31301519
- [Background] Rodriguez-Manas L, Fried LP. Frailty in the clinical scenario. Lancet. 2015 Feb 14;385(9968):e7-e9. doi: 10.1016/S0140-6736(14)61595-6. Epub 2014 Nov 6. No abstract available. PMID 25468154
- [Background] Izquierdo M, Merchant RA, Morley JE, Anker SD, Aprahamian I, Arai H, Aubertin-Leheudre M, Bernabei R, Cadore EL, Cesari M, Chen LK, de Souto Barreto P, Duque G, Ferrucci L, Fielding RA, Garcia-Hermoso A, Gutierrez-Robledo LM, Harridge SDR, Kirk B, Kritchevsky S, Landi F, Lazarus N, Martin FC, Marzetti E, Pahor M, Ramirez-Velez R, Rodriguez-Manas L, Rolland Y, Ruiz JG, Theou O, Villareal DT, Waters DL, Won Won C, Woo J, Vellas B, Fiatarone Singh M. International Exercise Recommendations in Older Adults (ICFSR): Expert Consensus Guidelines. J Nutr Health Aging. 2021;25(7):824-853. doi: 10.1007/s12603-021-1665-8. PMID 34409961
- See also: Projeto VIVIFRAIL — http://vivifrail.com
- See also: Tiecker, 2021 — http://tede2.pucrs.br/tede2/bitstream/tede/9693/2/TIECKER_ANA_PAULA_DIS.pdf